CLINICAL TRIAL: NCT04109183
Title: A Dose-exploratory Clinical Study of Azvudine Tablets in Patients Who Have Not Received Anti-HIV treatment--a Multicenter, Randomized, Double-blind, Double-simulation, Positive Control Trial
Brief Title: A Drug Safety and Dose-exploratory Clinical Study of Azvudine Tablets in Patients Who Have Not Received Anti-HIV Treatment
Acronym: FNC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Collaborators: Beijing YouAn Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Ditan Hospital (Other); Guangzhou 8th People's Hospital (Other); The Sixth People's Hospital of Zhengzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GQ-FNC-201
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: AIDS
Keywords: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: a multicenter, randomized, double-blind, double-simulation, positive control trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This experiment used a block randomization method, and each research center competed for inclusion. The SAS software (9.3 or above) was used to generate a random table and the corresponding treatment group for the random table. The clinical trial electronic central stochastic system (DAS for IWRS) was used to assign random numbers.Blind bottom sealed preservation, respectively sealed by the sponsor and clinical research unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Comparator: FNC 2 mg+ TDF+EFV (Experimental)
  Interventions: Drug: The subjects were randomized to the treatment group of 3TC or different doses of FNC. The background drugs were EFV and TDF.
- Active Comparator: FNC 3 mg+ TDF+EFV (Experimental)
  Interventions: Drug: The subjects were randomized to the treatment group of 3TC or different doses of FNC. The background drugs were EFV and TDF.
- Active Comparator: FNC 4 mg+ TDF+EFV (Experimental)
  Interventions: Drug: The subjects were randomized to the treatment group of 3TC or different doses of FNC. The background drugs were EFV and TDF.
- Postive Comparator: 3TC+ TDF+EFV (Experimental)
  Interventions: Drug: The subjects were randomized to the treatment group of 3TC or different doses of FNC. The background drugs were EFV and TDF.

INTERVENTIONS:
Drug: The subjects were randomized to the treatment group of 3TC or different doses of FNC. The background drugs were EFV and TDF. — The subjects were randomized to the treatment group of 3TC or different doses of FNC. The background drugs were EFV and TDF.

SUMMARY:
The primary objective of this trial was to evaluate the safety and preliminary evaluation of Azvudine tablets (FNC) in combination with reverse transcriptase inhibitors therapy in treatment-naive patients with HIV infection.; the secondary objective is to explore the effective dose of clinical use of Azvudine (FNC) tablets .

DETAILED DESCRIPTION:
Azvudine (FNC), a new class I drug with independent intellectual property rights, is a novel nucleoside reverse transcriptase inhibitor with good inhibitory activity against HIV-1 and obtained the National Medical Products Administration(NMPA) approved for clinical research.

In this trial, 172 patients who had not received anti-HIV treatment were enrolled, including FNC4mg group, FNC3mg group, FNC2mg group, and 3TC control group, 43 cases, 5 research centers, and each research center was simultaneously engaged and competing. The enrolled subjects underwent 7 visits including baseline visits, and HIV -1RNA and CD4 cell counts were tested and statistically analyzed for each visit.

ELIGIBILITY:
Inclusion Criteria:

1.18-65 years old, regardless of gender; 2.Confirmed HIV positive with a report; 3.Have not received anti-hiv antiviral treatment; 4.HIV viral load ≥1000 copies/mL; 5.Who have no recent family planning and agree to take effective non-drug contraceptive measures during the trial period and within 3 months after the end of administration; 6.The subjects could fully understand the purpose, nature, method and possible adverse reactions of the test, and voluntarily participate in and sign the informed consent.

Exclusion Criteria:

1. Patients who have received anti-HIV treatment;
2. Suffering from a serious opportunistic infection or opportunistic tumor;
3. Abnormal blood routine examination (white blood cells <3 × 109 / L, hemoglobin <90g / L, neutrophils <1.5 × 109 / L, platelets <75 × 109 / L);
4. Have a definite liver disease (hepatitis B surface antigen/HCV antibody positive), or abnormal liver function test (alanine aminotransferase and/or aspartate aminotransferase exceeds the upper limit of normal value by 3 times, or total bilirubin exceeds the upper limit of normal value 2 times);
5. Renal insufficiency (glomerular filtration rate <70ml/min, or creatinine above the upper limit of normal);
6. Now suffering from more serious chronic diseases, metabolic diseases (such as diabetes), neurological and psychiatric diseases;
7. Has suffered from pancreatitis;
8. Women during pregnancy and lactation;
9. allergic constitution or known to be allergic to the pharmaceutical ingredients and the basic drugs prescribed in this program;
10. Suspect or determine the history of alcohol and drug abuse;
11. Participated in other drug clinical trials (excluding Chinese medicine) within the first three months of screening;
12. Other factors that are not suitable for entering the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of azivudine tablet (FNC) combined with reverse transcriptase inhibitor therapy without anti-hiv treatment. | At 48 weeks
  Number of subjects with HIV viral load < 50copies/ml after treatment
Preliminary evaluation of the efficacy of azivudine tablets (FNC) combined with reverse transcriptase inhibitors in the treatment of patients who have not received anti-hiv treatment. | At 48 weeks
  Number of subjects with HIV viral load < 50copies/ml after treatment

SECONDARY OUTCOMES:
To explore the effective dose of azivudine tablet (FNC) in clinic | At 48 weeks
  Changes in HIV load logarithm before and after treatment, including the number of subjects whose HIV load level decreased by ≥1log from baseline before and after treatment;CD4 cell count before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing YouAn Hospital, Capital Medical University., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No